CLINICAL TRIAL: NCT01485965
Title: A Phase 1b, Open-label, Parallel-group Study in Subjects With Huntington Disease to Assess the Safety, Tolerability, and Fed/Fasted Pharmacokinetics of Repeated Oral Doses of SEN0014196
Brief Title: A Open-label Food Effect Study With SEN0014196 in Subjects With Huntington Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Siena Biotech S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S015-007
Record Dates: First submitted 2011-11-29; First posted 2011-12-06 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Huntington's Disease
Keywords: Huntington Disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Chorea; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Genetic Diseases, Inborn; Cognition Disorders; Mental Disorders
MeSH Terms: conditions — Huntington Disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Chorea; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Genetic Diseases, Inborn; Cognition Disorders; Mental Disorders | interventions — 6-chloro-2,3,4,9-tetrahydro-1H-carbazole-1-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted condition (Experimental): Subjects in the Fasted group will take study drug after an overnight fast (since at least midnight). Additionally, on PK assessment days, no food will be allowed for at least 4 hours after study drug administration.
  Interventions: Drug: SEN0014196
- Fed condition (Experimental): Subjects in the Fed group will take study drug within 30 minutes after starting breakfast; these subjects will otherwise maintain their normal eating schedule.
  Interventions: Drug: SEN0014196

INTERVENTIONS:
Drug: SEN0014196 — 100 mg, immediate release tablets, once daily administration

SUMMARY:
The primary purpose of this study is to assess the effect of food upon the pharmacokinetics (PK) of SEN0014196 in subjects with Huntington disease (HD).

DETAILED DESCRIPTION:
In addition to the pharmacokinetic endpoints, the study will assess the safety and tolerability of 100 mg once daily (qd) doses of SEN0014196 over 14 days in subjects with HD and explore potential biomarkers for use in subsequent Phase 2/3 studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with early to mid HD, i.e., genetically confirmed HD (cytosine, adenine, guanine [CAG] codon repeat length ≥ 36), motor signs of HD, and a Total Functional Capacity Subscale Score (TFC) ≥ 7
* Body mass index between 18 and 31 kg/m2 inclusive
* All subjects must have a body weight greater than 50 kg
* Female subjects must be surgically sterile, postmenopausal, or willing to practice a highly effective method of contraception. All female participants must be nonlactating and nonpregnant. Male subjects must agree to use a reliable method of birth control during the study and for 3 months after the last dose of study drug.
* Capable of providing informed consent
* MMSE ≥24
* Subjects must have a live-in competent observer

Exclusion Criteria:

* Participation in a study or received an investigational drug within 30 days of the Baseline Visit
* Any prior or concomitant use of compounds suspected of interfering with protein acetylation
* Any concomitant use of medications that are known inhibitors of CYP450 enzymes or substrates of CYP1A2 at the time of enrollment
* Suicide risk, as determined by meeting either of the following criteria: a) a suicide attempt within the past year or suicidal ideation within 60 days of the Screening Visit; b) Significant risk of suicide, as judged by the Investigator
* Subjects with MMSE < 24
* Subjects with presence of clinically significant psychosis and/or confusional states, in the opinion of the Investigator
* Subjects with clinically significant laboratory or ECG abnormalities at Screening or Baseline
* Subjects with clinically relevant hematologic, hepatic, cardiac, or renal disease
* Subjects with a current or past (within the last 12 months) history of epilepsy or seizures
* A medical history of infection with human immunodeficiency virus, hepatitis C, and/or hepatitis B
* Subjects with a history of substance abuse within the past 12 months
* Female subjects who are pregnant or breastfeeding
* Known allergy to any ingredient in the study drug
* A history of malignancy of any type within 2 years prior to Screening. A history of surgically-excised nonmelanoma skin cancers is permitted.
* Any relevant condition, behavior, laboratory value, or concomitant medication which, in the opinion of the Investigator, makes the subject unsuitable for entry into the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of food on the repeated dose pharmacokinetics of SEN0014196 at 100 mg once daily in subjects with Huntington's disease | 14 Days
  The effect of food on the PK of SEN0014196 will be evaluated for the following parameters: maximum observed plasma concentration (Cmax), time of maximum observed plasma concentration(tmax), AUC from time zero to the length of the dosing interval (tau) (AUC0-τ), AUC from time zero to the last quantifiable concentration (AUC0-last), AUC from time zero to infinity (AUC0-∞), terminal elimination half-life (t1/2), and terminal elimination rate constant (λz).

SECONDARY OUTCOMES:
Pharmacodynamics | 14 Days
  The following PD biomarkers will be assessed: soluble huntingtin levels and huntingtin acetylation status (by enzyme-linked immunosorbent assay [ELISA] and liquid chromatography-tandem mass spectrometry [LC-MS/MS]).
To determine the safety and tolerability of repeated doses of SEN0014196 at 100 mg once daily in subjects with Huntington's disease | 14 Days
  Safety assessments include: AEs, ECGs, vital signs, body weight and height, clinical laboratory evaluations (serum biochemistry and hematology), urinalysis, physical and neurological examinations, C-SSRS, and UHDRS.

CONTACTS AND LOCATIONS:
Overall Officials: Francis O Walker, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - University of California San Diego, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - Washington University, St Louis, Missouri
  - University of Rochester, Rocherster, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas